CLINICAL TRIAL: NCT06014372
Title: A Prospective, Single-center, Multi-cohort Study of Envolimab Monotherapy or Envafolimab in Combination With CAPEOX as Neoadjuvant Therapy for Locally Advanced Colorectal Cancer.
Brief Title: Envafolimab Monotherapy or Envafolimab + CAPEOX as Neoadjuvant Therapy for Locally Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhen-Hai Lu, Prof., Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-FXY-256-Department of CRC
Record Dates: First submitted 2023-08-23; First posted 2023-08-28 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Colon Cancer; Neoadjuvant Therapy; Immunotherapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — envafolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Envafolimab Group (Experimental): Patients diagnosed with colon cancer, with T stage determined as 3-4 based on enhanced MR imaging, or with any T stage accompanied by imaging findings suggestive of lymph node metastasis, and excluding patients with distant metastasis, who are confirmed to have microsatellite instability-high (MSI-H)/deficient mismatch repair (dMMR) colon cancer, will be enrolled in Group A
  Interventions: Drug: Envafolimab
- Envafolimab+CAPEOX Group (Active Comparator): Patients diagnosed with colon adenocarcinoma, with T stage determined as 3-4 based on enhanced MR imaging, or with any T stage accompanied by imaging findings suggestive of lymph node metastasis, and excluding patients with distant metastasis, who are confirmed to have microsatellite stable (MSS)/proficient mismatch repair (pMMR) colon cancer, will be enrolled in Group B.
  Interventions: Drug: Envafolimab; Drug: CAPEOX

INTERVENTIONS:
Drug: Envafolimab — Upon confirming eligibility based on inclusion criteria and obtaining signed informed consent, the patient will be administered Envafolimab at a dose of 300mg every 3 weeks (Q3W) for a total of 4 cycles, starting on Day 1.
Drug: CAPEOX — The neoadjuvant treatment regimen will consist of Oxaliplatin at a dose of 130mg/m2, administered intravenously over a period of more than 2 hours on Day 1, every 3 weeks; and Capecitabine at a dose of 1000mg/m2, orally, twice daily from Day 1 to Day 14, every 3 weeks, for a total of 4 cycles.
  Arms: Envafolimab+CAPEOX Group

SUMMARY:
There exists substantial evidence suggesting that patients diagnosed with MSI-H/dMMR colorectal cancer can derive benefits from immunotherapy in the management of advanced colorectal cancer. In cases of locally advanced colorectal cancer exhibiting microsatellite instability (dMMR/MSI-H), patients exhibit low responsiveness to neoadjuvant chemotherapy, resulting in minimal rates of complete tumor remission and downstaging. Nevertheless, initial exploratory studies, characterized by modest sample sizes, reveal a favorable therapeutic effect of neoadjuvant immunotherapy in this particular patient population. Envafolimab monoclonal antibody, the first PD-L1 antibody developed and manufactured in China, possesses noteworthy practical and societal value in the context of exploratory clinical research on neoadjuvant immunotherapy for locally advanced MSI-H/dMMR colorectal cancer patients. The objective of this study is to evaluate the safety and efficacy of envafolimab monoclonal antibody (PD-L1) as neoadjuvant therapy for locally advanced MSI-H/dMMR colorectal cancer through a prospective, multi-cohort phase II clinical trial. Additionally, this study aims to investigate the effectiveness and safety of envafolimab monoclonal antibody in combination with CAPEOX as a neoadjuvant treatment regimen for locally advanced pMMR colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmed rectal cancer
* Clinical stage T3-4 or T any N1
* With or without MRF positivity, with or without EMVI positivity
* R0 resection is estimated
* Age ranged from 18 to 70

Exclusion Criteria:

* Clinical stage T1-2 N0
* Distance metastasis
* Multiple primary tumor
* Cachexy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of pCR | Time Frame: One week after surgery
  rate of pathological complete remission

SECONDARY OUTCOMES:
DFS | 3 years
  Disease free survival

OTHER OUTCOMES:
OS | 5 years
  O Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China